CLINICAL TRIAL: NCT06977477
Title: Managing Congestion in Heart Failure: Pressure- and Volume- Based. A Mechanistic Study in Patients With HFpEF (MAGIC-HF)
Brief Title: Managing Congestion in Heart Failure: A Mechanistic Study in Patients With HFpEF
Acronym: MAGIC-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Otto-von-Guericke University Magdeburg (Other)
Responsible Party: Principal Investigator, Tarek Bekfani, MD, MSc (Oxon.), FESC, FHFA, Otto-von-Guericke University Magdeburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 30/24
Record Dates: First submitted 2025-05-09; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Remote Monitoring in Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with HFpEF Remotely Monitored for Congestion and Volume Management (Other): Patients with HFpEF will undergo remote monitoring for congestion management using daily measurements of pulmonary artery pressure via CardioMEMSTM and body water volumes through a smart scale using bioelectrical impedance analysis (BIA). Body water volume will be tracked in different segments (arms, legs, trunk), alongside pulmonary pressure, to explore the mechanisms of congestion and describe its varied phenotypes in HFpEF patients. This intervention aims to optimize fluid balance management and improve clinical outcomes.
  Interventions: Other: Remote Monitoring for Congestion Management in HFpEF Patients

INTERVENTIONS:
Other: Remote Monitoring for Congestion Management in HFpEF Patients — All patients will undergo baseline tests, including echocardiography (left ventricular ejection fraction, E/e', left atrial volume index, left atrial strain analysis, left ventricular mass index, tricuspid annular plane systolic excursion, right ventricular strain, inferior vena cava index) and blood tests (NT-proBNP, creatinine, GFR, sST2, CA 125, bio-ADM, ALAT, ASAT, complete blood count, and hsCRP). Evaluation of extracellular and total body water volumes in the arms, legs, and trunk will be conducted using the Body Water Scale InBody (South Korea) and daily monitoring of pulmonary pressure through CardioMEMSTM. Bioelectrical impedance analysis (BIA) will be used to assess volume. Additional blood tests will be conducted at weeks 2, 6, 12, and at the final visit, with a focus on NT-proBNP, creatinine, GFR, ALAT, ASAT, hemoglobin, hematocrit, hsCRP, sST2, CA 125, and bio-ADM. At the final visit, a complete set of tests will be repeated to assess overall health and response to the int

SUMMARY:
The goal of this clinical trial (MAGIC-HF) is to understand whether daily remote monitoring of pulmonary artery pressure using the CardioMEMS™ device and body water levels using a smart scale can improve the management of congestion in people with heart failure with preserved ejection fraction (HFpEF). Participants who already have an indication for remote monitoring with CardioMEMS™ (A sensor to be implanted in the pulmonary artery in a minimal invasive procedure) will be enrolled. Every day, patients will measure their pulmonary pressure using CardioMEMS and assess the amount of water in different parts of the body, including the arms, legs, and trunk using the scale BWA ON. The measurements will take about 2 minutes each. Over a period of six months, researchers will monitor these measurements along with regular blood tests to observe changes in heart and kidney function by monitoring biomarkers reflecting the function of these organs.

Managing fluid buildup (congestion) is a major challenge in people with heart failure, and current methods based on clinical signs are not always reliable. Recent research suggests that congestion in heart failure is not only related to pressure but also to changes in fluid volume, and that better monitoring could help tailor treatments more effectively. By combining pressure and volume data, this study aims to help reach a more balanced fluid state (euvolemia) in participants, which could reduce hospital readmissions and improve overall outcomes. In addition, the study seeks to identify different types, or phenotypes, of congestion based on pressure and volume profiles, which could guide more personalized care in the future.

This study is important because it addresses an urgent need to improve the early detection and management of congestion in heart failure. It also explores new approaches that could lead to better understanding and treatment of this complex condition, especially in patients with preserved ejection fraction who often have fewer treatment options.

DETAILED DESCRIPTION:
Heart failure with preserved ejection fraction (HFpEF) remains a major clinical challenge, with high hospitalization and readmission rates that contribute to substantial healthcare costs. Achieving and maintaining euvolemia is a key goal in the management of heart failure (HF), but current methods of monitoring congestion are suboptimal. Clinical signs and symptoms often occur late and are neither sensitive nor specific for detecting early decompensation. Furthermore, traditional reliance on pressure measurements alone, such as pulmonary artery pressures, has been questioned, since elevated pressure may coexist with euvolemia or hypovolemia.

The MAGIC-HF study is a prospective, mechanistic, multi centre, remote monitoring (RM) study aiming to explore the combined use of pressure- and volume-based monitoring to improve congestion management in patients with HFpEF and to better understand the relation pressure-volume in this group of patients. This study will evaluate the daily measurements of pulmonary artery pressure, collected via the CardioMEMS™ device, in conjunction with extracellular and total body water assessments obtained through a segmental bioelectrical impedance smart scale (BWA device).

Participants enrolled in the study will have an indication for CardioMEMS™ monitoring and will undergo continuous daily assessments over a 6-month follow-up period. These measurements will focus on changes in pulmonary pressure and body fluid distribution across upper extremities, lower extremities, and trunk compartments. The hypothesis is that combining pressure and volume data will allow better detection and management of congestion, reaching a euvolemic state more effectively, and ultimately improving important biomarkers such as NT-proBNP and renal function.

Baseline evaluations will include a comprehensive echocardiographic assessment: laboratory analyses (NT-proBNP, creatinine, GFR, sST2, CA-125, bio-ADM, ALAT, ASAT, complete blood count, hsCRP). Daily remote monitoring will involve CardioMEMS™ pressure recordings and smart scale assessments. Additional blood tests will be collected at days 14, 42, 90, and at the final visit.

The study aims to characterize different congestion phenotypes based on pressure-volume relationships, such as elevated pressure with hypervolemia, euvolemia, or hypovolemia. Understanding these subgroups may allow tailored management strategies. This could challenge current treatment paradigms, particularly the routine use of diuretics based solely on pressure readings.

The primary focus will be an exploratory analysis of changes in NT-proBNP levels, glomerular filtration rate (GFR), and the proportion of participants presenting with discordant pressure and volume statuses. NT-proBNP will be adjusted for BMI following formulas used in previous trials like GUIDE-HF.

Overall, MAGIC-HF seeks to expand knowledge of congestion mechanisms in HFpEF, inform clinical practice about more precise management of congestion, and potentially lead to improved clinical outcomes through more individualized and physiologically guided therapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patients with HFpEF, who are hospitalized for acute decompensated heart failure and require treatment with intravenous (IV) diuretics.
* Signed informed consent.

Exclusion Criteria:

* Patients admitted with cardiogenic shock and/or those who required inotropic or vasopressor support.
* Had a history of cardiac transplantation or ventricular assist device (VAD) implantation.
* Had any implanted cardiac device (pacemaker, ICD, CRT-D.
* Had chronic kidney disease with creatinine clearance < 20 ml/min.
* Had recent acute MI or CABG within 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
The Percentage of Patients with Elevated Pulmonary Pressure but Hypo- or Euvolemic and vice versa at 6 Months | 6 months
  describing the phenotypes of different volume-pressure patterns and the thus better understanding the mechanism of congestion development.
Change from Baseline in GFR (mL/min/1.73m2) | 6 months
  safety Outcome

SECONDARY OUTCOMES:
Change from Baseline of NT-proBNP Levels (pg/ml) | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Otto von Guericke University, Faculty of Medicine, Magdeburg, Saxony-Anhalt, Germany

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2024-12-17): https://cdn.clinicaltrials.gov/large-docs/77/NCT06977477/Prot_000.pdf